CLINICAL TRIAL: NCT03967912
Title: Mobility and Vitality Lifestyle Program-Caregivers
Brief Title: MOVE UP Lifestyle Intervention for Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven M. Albert, Professor and Chair, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY18110005; U48DP005001 (NIH)
Record Dates: First submitted 2019-05-24; First posted 2019-05-30 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Body Weight; Healthy Diet; Physical Activity; Health Behavior; Healthy Aging
MeSH Terms: conditions — Body Weight; Motor Activity; Health Behavior

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Implementation research for adapted effective intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOVE UP for Caregivers (Experimental): 12-week lifestyle intervention focusing on diet and activity
  Interventions: Behavioral: MOVE UP

INTERVENTIONS:
Behavioral: MOVE UP — Each of the 12 group sessions will focus on incremental behavioral strategies for maintaining healthy eating, activity, and weight loss.behaviors. Body weight will be measured in-person session and participants will also to measure their body weight on their in Session 3, participants are given physical activity goal of 10 minutes/day, 50 minutes/week. The goal is raised by 5 minutes/day, 25 minutes/week every other session, the final goal being 30 minutes/day, 150 minutes/week. All subjects will be recommended to engage in an energy restricted dietary intervention that evidence demonstrates has effectively reduced body weight by 5-7% within the initial 4 months of the intervention. This will include reducing energy intake to 1200 to 1800 kcal/d based on initial body weight (<200 pounds = 1200 kcal/d; 200 to 250 pounds = 1500 kcal/d; >250 pounds = 1800 kcal/d).

SUMMARY:
In prior research the Mobility and Vitality Lifestyle Program for healthy aging and weight management (MOVE UP) was effective in producing a mean loss of >= 5% body weight, with increased physical activity and reduced fatigue. This research will pilot a modified and streamlined version to see if it will be similarly effective for caregivers of family members or friends who have dementia, physical and/or developmental issues, or health problems.

DETAILED DESCRIPTION:
The investigators aim to test the feasibility of delivery of a modified and streamlined lifestyle program in volunteer community settings and to provide pilot data to inform the design of future randomized controlled trials that may improve physical and mental health in older adults (50-75) who are providing care for a family member or friend who has dementia, physical and/or developmental issues, or health problems. Current objectives include:

1 . Adapt and pilot the previously studied 32-session, 13-month MOVE UP intervention to a streamlined 12-session (4-month) community-based translational behavioral weight management program. The pilot program will be delivered by a staff interventionist.

2. Implement and evaluate the program's impact on weight and healthy lifestyle changes, including physical performance outcomes, at 2 sites, each with at least 6 eligible obese and caregiving adults ages 50-75 years old.

ELIGIBILITY:
Inclusion Criteria:

1. 50-75 years of age
2. BMI >=27.0, but <45.0
3. Able to consent for participation and data collection.
4. Medical clearance from physician/health care provider before session 2 in program.
5. Ability to walk with or without assistive device.
6. Acting as a caregiver to someone with dementia, a serious illness, and/or a developmental or physical disability.

Exclusion Criteria:

1. Past MOVE UP participant.
2. If weight loss in the past year is >=10% body weight.
3. Use of wheelchair; participant must be willing and able to increase physical activity.
4. Uncontrolled diabetes mellitus (FBS > 30 & A1C > 11%); to be assessed by physician on medical release.
5. Uncontrolled hypertension (SBP > 180/110) %); to be assessed by physician on medical release.
6. Recent overnight hospitalization (past 6 months).
7. Active treatment for cancer (including melanoma).
8. Significant visual or hearing impairment.
9. Significant cognitive disorder/relevant and significant psychiatric disorder (to be assessed on medical release).
10. Inability to communicate in English/lack of translator.
11. Currently enrolled in another research study that could impact study outcomes or interfere with either study. Exclude if less than 12 months post-graduation from previously enrolled study.
12. Currently enrolled in a weight loss program, such as Weight Watchers.
13. Inability or unwillingness to attend the majority of sessions.
14. In the past year, participating in (other) ways of losing weight, such as bariatric surgery, prescription medications, or non-surgical interventions (reviewed by investigators).
15. Unable to obtain medical clearance by session 2.
16. Not acting as a caregiver.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Body weight change from Baseline to 4 months | 4 months
  Number of participants with at least a 5% decrease in body weight from baseline at 4 months

SECONDARY OUTCOMES:
Change in objectively measured physical function from Baseline to 4 months | 4 months
  Observed performance measure using SPPB. Scores range from 0 (worst performance) to 12 (best performance)
Change in physical function from Baseline to 4 months | 4 months
  Self-reports using CHAMPS. Score range is 0- 793, with higher scores indicating greater physical activity.
Change in psychosocial measures from Baseline to 4 months | 4 months
  Self-report using CES-D. Score range 0-60, in which higher scores suggest a greater presence of depressive symptoms.
Changes in physical, mental, and social health | 4 months
  Self-report using PROMIS ® (Patient-Reported Outcomes Measurement Information System), which is a set of person-centered measures that evaluates physical, mental, and social health. The PROMIS-29 consists of self-report items from seven domains (Depression, Anxiety, Physical Function, Pain Interference, Fatigue, Sleep Disturbance, and Ability to Participate in Social Roles and Activities). Summed scores from each domain can be converted into a T-score using a table provided by test developers. The table rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A score of 50 is the average for the United States general population, and a person with a T-score of 40 is one SD below the mean. For this exploratory measure we are interested to establish effect sizes for MOVE UP, that is, how much of a change in T score is on average associated with the MOVE UP lifestyle intervention.
Changes in caregiver burden | 4 months
  Self-report using Short Form Zarit Burden Interview (ZBI-12). Score range 0-48, in which higher scores indicate a greater burden.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Albert, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Prevention Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venditti EM, Zgibor JC, Vander Bilt J, Kieffer LA, Boudreau RM, Burke LE, Glynn NW, Jakicic JM, Smith KJ, Semler LN, Rager JR, Albert SM, Newman AB. Mobility and Vitality Lifestyle Program (MOVE UP): A Community Health Worker Intervention for Older Adults With Obesity to Improve Weight, Health, and Physical Function. Innov Aging. 2018 Jun 18;2(2):igy012. doi: 10.1093/geroni/igy012. eCollection 2018 Jun. PMID 30480135

DOCUMENTS (1):
  • Informed Consent Form (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT03967912/ICF_000.pdf